CLINICAL TRIAL: NCT02544035
Title: Determining Age Appropriateness of Children's Products and Toys: An Interagency Agreement With the Consumer Product Safety Commission
Brief Title: Determining Age Appropriateness of Children's Products and Toys
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 999915196; 15-CH-N196 (Other: NIHCC)
Record Dates: First submitted 2015-09-05; First posted 2015-09-09 (Estimated); Results first posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2021-04-30

CONDITIONS: Healthy Volunteers Only
Keywords: Childhood Growth and Development; Development

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- 36-71 month-old Play Partner (Experimental): 36-71 month-olds (1.5-2 year olds)
  Interventions: Other: Play Partner
- 72-107 month-old Play Partner (Experimental): 72-107 month-olds (6-8 year-olds)
  Interventions: Other: Play Partner
- 12-18 month-old Toy Type (Experimental): 12-18 month-olds (1-1.5 year olds)
  Interventions: Other: Type of Toy
- 19-35 month-old Toy Type (Experimental): 19-35 month-olds (1.5-2 year-olds)
  Interventions: Other: Type of Toy
- 36-71 month-old Toy Type (Experimental): 36-71 month-olds (3-5 year-olds)
  Interventions: Other: Type of Toy
- 72-107 month-old Toy Type (Experimental): 72-107 month-olds (6-8 year-olds)
  Interventions: Other: Type of Toy
- 12-18 month-old Play Partner (Experimental): 12-18 month-olds (1-1.5 year olds)
  Interventions: Other: Play Partner
- 19-35 month-old Play Partner (Experimental): 19-35 month-olds (1.5-2 year olds)
  Interventions: Other: Play Partner

INTERVENTIONS:
Other: Type of Toy — Children will be presented with one of three (counterbalanced) toys targeted for their age group. When presented, each target toy will be paired with two additional toys from the same toy category;
  Arms: 12-18 month-old Toy Type; 19-35 month-old Toy Type; 36-71 month-old Toy Type; 72-107 month-old Toy Type
Other: Play Partner — Each child will first play alone then play with parent.
  Arms: 12-18 month-old Play Partner; 19-35 month-old Play Partner; 36-71 month-old Play Partner; 72-107 month-old Play Partner

SUMMARY:
Background:

Play during childhood is an important part of healthy development, and children can learn many things when they play. Much of the time that children spend playing is with toys. However, children at different ages need different types of toys to engage in healthy play.

Understanding children s play with toys is important to the National Institute of Child Health and Human Development (NICHD), and to the U.S. Consumer Product Safety Commission (CPSC). The CPSC rates toys that are currently available in the United States for children for age appropriateness. NICHD will share the findings of this study with CPSC to aid in their toy rating process.

Objective:

To categorize traditional and contemporary children s products and toys into age appropriate groups.

Eligibility:

Healthy children 6 months to 12 years old.

Their parents.

Design:

Participants will be screened with a phone call with the parents.

Participants will complete surveys online or on paper, and by phone. These will ask about demographic facts, behavior, thoughts on parenting and toys, and child development.

Participants will have 1 study visit. The child will play with toys by himself or herself. Then they will play with their parent. A researcher will observe. The sessions will be videotaped.

Children will share their thoughts about the toys by pointing at a smiley face scale.

Parents will fill out a short survey. Then can choose to participate in a 1-hour focus group.

DETAILED DESCRIPTION:
The proposed project is the outcome of an interagency agreement (IAG; #CPSC-I-14-0016) between the Consumer Product Safety Commission (CPSC) of the United States and the Child and Family Research Section (CFRS) within NICHD DIR. At the CPSC, the Division of Human Factors (ESHF) examines products and toys for U.S. children and determines the appropriate age of their potential users based on a set of Guidelines last revised in 2002. Due to the outdated nature of the 2002 Guidelines, the CFRS is charged with revising this rulebook after conducting an empirical research project to inform these amendments. The goal of the current study is to categorize traditional and contemporary children s products and toys into age appropriate groups and use this information to rewrite the Guidelines for efficient CPSC use.

Participants will be 360 parent-child dyads from 6 months to 12 years of age. We will recruit equal numbers of boys and girls from each of the following six developmentally determined and CPSC approved age groups: 6-11 mos, 12-18 mos, 19-35 mos, 36-71 mos (3-5 years), 72-107 mos (6-8 years), and 108-144 mos (9-12 years). Participants will be tested at the CFRS once parental consent and child assent have been obtained.

Each child will receive one of three counterbalanced children s products or toys that are targeted to their age group from 6 of the 9 following categories: (1) Building or Construction (e.g., blocks, interlocking building materials), (2) Exploratory (e.g., clay, sand toys), (3) Games & Puzzles, (4) Instructional Toys (e.g., books, science kits), (5) Sports, Recreation, & Outdoor, (6) Imaginative Play (e.g., puppets, dolls, dress up materials), (7) Small Wheeled Vehicles (e.g., car toys), (8) Arts and Crafts, and (9) Musical Toys (e.g., musical instruments). Children will also receive one of three (counterbalanced) children s products or toys from each of the categories aimed at the age group below their age as well as another from each of the categories aimed at the age group older than their age. Each child will first play alone and then play with a parent. Different sets of toys will be presented when children switch from playing alone to playing in a dyad.

Parents will provide information about their socioeconomic status and demographics. They will also complete the Vineland Adaptive Behavior Scales (i.e., an instrument assessing the child s socialization, motor, communication, and daily living skills) and an age-appropriate instrument that assesses the child s temperament. They will provide information about toys that are already in their home. Some parents may be invited to take part in a more in-depth qualitative focus group interview about children s toys. All play sessions will be video recorded and will be scored for relevant behaviors.

We will examine differences in play with toys from the three age groups that are chronologically adjacent (i.e., to determine differences in outcomes for a given age group with age-appropriate toys compared to toys of the same category from the next youngest and next oldest age groupings). Our outcome measures include the following: (1) Complexity of play, (2) Parts and features of toys used by the child, (3) Duration of time spent with each toy, (4) Preference for the toys, and (5) Number of times and duration the child solicits the parent s involvement during play.

This observational study of children fits well with the CFRS program of research and the mission of the NICHD DIR. We will investigate children s interactions with toys that surround children in their natural environment, as well as study how parents moderate child play behavior. Observing and quantifying behaviors during play will allow us to have a richer understanding of social and cognitive growth during different stages of child development in the context of toy play with parents and will form an empirical basis for revising the 2002 CPSC Guidelines in light of changes in the last decade and a half in the toy industry.

The cost impact for this project is minimal. All necessary testing facilities are already available at the CFRS. Funding for additional staff needed to work with participants, subject reimbursement, and supplies to carry out the project is allocated through the IAG.

ELIGIBILITY:
* INCLUSION CRITERIA:

All children between the ages of 6 months to 12 years of age who are typically developing and born of a full term pregnancy if under 24 months of age, healthy, and English speaking are eligible for inclusion in the study. Typically developing children would not have any diagnosed congenital conditions, developmental delay or disability, dyslexia, PDD, ADD, ADHD, or ASD. In addition, we will only enroll subjects if they are from a racial and ethnic group that is still needed to ensure the diversity and representative nature of our sample as set forth in the Planned Enrollment Form. These are the initial screening criteria that will be used.

EXCLUSION CRITERIA:

* Children outside of the 6 month-12 year age range: These years cover early life and are the ages of interest for children s play and are of central significance to the Consumer Product Safety Commission s goals.
* Families not fluent in English: Fluency in English is essential for parents to be able to fill out surveys. Families also need to be fluent in English so that they can comprehend verbal directions given by the experimenter during the testing session. If we included people who were not fluent in English, we would need many additional staff members who speak the multitude of languages of the diverse population of the Washington, D.C metro area to work with participants during the testing session and code the videos after the testing session is complete.
* Children who are sick, not typically developing, born premature (if they are under 24 months of age), blind, or deaf: We must recruit a healthy sample of typically developing children born in a full term pregnancy (if they are under 24 months of age) who are not blind or deaf for this project to remove any potential confounds that atypical conditions may have on children s play. Typically developing children would not have any diagnosed congenital conditions, developmental delay or disability, dyslexia, PDD, ADD, ADHD, or ASD. Including other populations such as deaf or blind children would require a different experimental set up, stimulus toys, and resources (i.e., someone who could convert our surveys to American Sign Language or Braille and could code the videos for the parent child behaviors during those sessions).
* Children who are not adding to the ethnic and racial diversity of the sample: The goal of our study is to recruit a sample of subjects who are racially and ethnically diverse. By making this diverse sample a priority, we hope that our results will be applicable to the diverse populations residing within the United States. To keep with this goal of a diverse and representative sample of children, we may have to exclude some families if we have already reached the quota of families from that particular racial or ethnic group.

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 486 (Actual)
Dates: Start 2015-09-05; Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diane L Putnick, Ph.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institute of Child Health and Human Development (NICHD), Bethesda, Maryland, United States

REFERENCES:
- [Background] Bornstein MH, Haynes OM, O'Reilly AW, Painter KM. Solitary and collaborative pretense play in early childhood: sources of individual variation in the development of representational competence. Child Dev. 1996 Dec;67(6):2910-29. PMID 9071765
- [Result] Richards MN, Putnick DL, Bradley LP, Lang KM, Little TD, Suwalsky JTD, Bornstein MH. Children's Utilization of Toys is Moderated by Age-Appropriateness, Toy Category, and Child Age. Appl Dev Sci. 2022;26(1):192-205. doi: 10.1080/10888691.2020.1760868. Epub 2020 May 19. PMID 35110960
- [Result] Richards MN, Putnick DL, Bornstein MH. Toy Buying Today: Considerations, Information Seeking, and Thoughts about Manufacturer Suggested Age. J Appl Dev Psychol. 2020 May-Jun;68:101134. doi: 10.1016/j.appdev.2020.101134. Epub 2020 Apr 8. PMID 32405125

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 12-18 Month-old Toy Type | 19-35 Month-old Toy Type | 36-71 Month-old Toy Type | 72-107 Month-old Toy Type | 12-18 Month-old Play Partner | 19-35 Month-old Play Partner | 36-71 Month-old Play Partner | 72-107 Month-old Play Partner
Started | 60 | 61 | 62 | 60 | 60 | 61 | 62 | 60
Completed | 60 | 61 | 62 | 60 | 60 | 61 | 62 | 60
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Children aged 6-11 months were dropped from inclusion because they were not reliably able to play with toys in pilot testing.
  Children aged 108-144 months were dropped from inclusion because few toys were identified as age appropriate for this group.
Groups:
- Total: Total of all reporting groups
Arm/Group | 12-18 Month-old Toy Type | 19-35 Month-old Toy Type | 36-71 Month-old Toy Type | 72-107 Month-old Toy Type | 12-18 Month-old Play Partner | 19-35 Month-old Play Partner | 36-71 Month-old Play Partner | 72-107 Month-old Play Partner | Total
Number analyzed (Participants) | 60 | 61 | 62 | 60 | 60 | 61 | 62 | 60 | 486
Age, Continuous [Mean (Standard Deviation); unit: months] | 15.34 (2.02) | 26.88 (4.96) | 54.16 (10.77) | 89.52 (11.42) | 15.34 (2.02) | 26.88 (4.96) | 54.16 (10.77) | 89.52 (11.42) | 46.46 (29.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 33 | 31 | 28 | 26 | 33 | 31 | 28 | 236
  Male | 34 | 28 | 31 | 32 | 34 | 28 | 31 | 32 | 250
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 6 | 8 | 5 | 3 | 6 | 8 | 44
  Not Hispanic or Latino | 55 | 58 | 56 | 52 | 55 | 58 | 56 | 52 | 442
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 8 | 4 | 4 | 4 | 8 | 4 | 4 | 40
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 5 | 4 | 8 | 4 | 5 | 4 | 8 | 42
  White | 40 | 41 | 42 | 36 | 40 | 41 | 42 | 36 | 318
  More than one race | 12 | 7 | 12 | 12 | 12 | 7 | 12 | 12 | 86
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 60 | 61 | 62 | 60 | 60 | 61 | 62 | 60 | 486

OUTCOME MEASURES:

1. Primary Outcome: Utilization of Toy
Description: Children's play with each of the toys was categorized as fully utilized (1) or not fully utilized (0) according to the intended use of each toy
Time Frame: 1 hour play session
Population: Child age by toy age appropriateness
Measure: Number; unit: Proportion
Arm/Group | 12-18 Month-old Toy Type | 19-35 Month-old Toy Type | 36-71 Month-old Toy Type | 72-107 Month-old Toy Type | 12-18 Month-old Play Partner | 19-35 Month-old Play Partner | 36-71 Month-old Play Partner | 72-107 Month-old Play Partner
Number analyzed (Participants) | 60 | 61 | 62 | 60 | 0 | 0 | 0 | 0
Proportion | .45 | .49 | .50 | .53 |  |  |  |

2. Secondary Outcome: Played With Toy
Description: We constructed a variable to indicate whether the child played with the toy (1) or did not play with the toy (0).
Time Frame: 1 hour play session
Measure: Number; unit: Proportion
Arm/Group | 12-18 Month-old Toy Type | 19-35 Month-old Toy Type | 36-71 Month-old Toy Type | 72-107 Month-old Toy Type
Number analyzed (Participants) | 60 | 61 | 62 | 60
Proportion | .67 | .61 | .62 | .65

3. Secondary Outcome: Duration of Toy Play
Description: Duration of time child plays with each toy
Time Frame: 1 hour play session
Reporting Status: Not Posted

4. Secondary Outcome: Preference for the Toy - Child-report
Description: Child preference for the toys based on child-report
Time Frame: 1 hour play session
Reporting Status: Not Posted

5. Secondary Outcome: Solicits to Parent Involvement
Description: Number of times child solicits parent involvement
Time Frame: 1 hour play session
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year 11 months
Description: Adverse events were defined consistent with the clinicaltrials.gov definitions.
Arm/Group | 12-18 Month-old Toy Type | 19-35 Month-old Toy Type | 36-71 Month-old Toy Type | 72-107 Month-old Toy Type | 12-18 Month-old Play Partner | 19-35 Month-old Play Partner | 36-71 Month-old Play Partner | 72-107 Month-old Play Partner
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/61 | 0/62 | 0/60 | 0/60 | 0/61 | 0/62 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/61 | 0/62 | 0/60 | 0/60 | 0/61 | 0/62 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/61 | 0/62 | 0/60 | 0/60 | 0/61 | 0/62 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-15): https://cdn.clinicaltrials.gov/large-docs/35/NCT02544035/Prot_SAP_000.pdf